CLINICAL TRIAL: NCT04081506
Title: Targeting the Optimal Mean Arterial Pressure in Hypoxic Ischemic Brain Injury After Cardiac Arrest
Acronym: CAMPING
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Myp Sekhon, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H16-00466-A015
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Individualized care
  Interventions: Other: Individualized perfusion targets
- Group B (No Intervention): Conventional care

INTERVENTIONS:
Other: Individualized perfusion targets — Targeting +/-5mmHg of the optimal mean arterial pressure
  Arms: Group A

SUMMARY:
Hypoxic ischemic brain injury (HIBI) is the ensuing brain injury after cardiac arrest and is the primary cause of adverse outcome. HIBI is caused by low oxygen delivery to the brain. The patient's blood pressure is primary determinant of oxygen delivery to the brain. International guidelines recommend maintaining uniform blood pressure targets in all patients, however, this 'one size fits all approach' fails to account for individual baseline differences between patient's blood pressures and extent of underlying disease. Recently, 'autoregulation monitoring', a novel brain monitoring technique, has emerged as a viable tool to identify patient specific blood pressures after brain injury. This personalized medicine approach of targeting patient specific blood pressure (MAPopt) is associated with improved outcome in traumatic brain injury. It has not been evaluated in HIBI after cardiac arrest.

Recently, I completed a first-in-human study demonstrating the ability to identify MAPopt in HIBI patients using neuromonitoring (microcatheters inserted into the brain tissue). The proposed study in this grant is to take the next step and investigate the changes in key brain physiologic variables (brain blood flow and oxygenation) before and after therapeutically targeting MAPopt in HIBI patients. This interventional study will serve as the basis to embark on a pilot randomized control trial of MAPopt targeted therapy versus standard of care in HIBI patients after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* We will include any patient 19 years or older who are admitted to the ICU following cardiac arrest with a post-resuscitation Glasgow Coma Scale of 8 or less.

  * Existing arterial line in situ as part of their clinical care.
  * Enrolled within 72 hours of their cardiac arrest
  * Patients must have had more than 20 consecutive minutes of spontaneous circulation following resuscitation
  * Duration of cardiac arrest greater than 10 minutes prior to return of spontaneous circulation. This is to ensure that we will not be placing intra-parenchymal bolts in patients who are likely to have a favourable neurological outcome regardless of monitoring.

Exclusion Criteria:

1. Coagulopathy (INR > 1.5, PTT > 40, Platelets < 100)
2. Cardiac catheterization procedure is anticipated within the next 7 days.
3. Current or anticipated use of anticoagulant or antiplatelet medication. Importantly, subcutaneous heparin or dalteparin for deep venous thrombosis prophylaxis may be used provided it is not administered 12 hours prior to insertion or removal of the bolt. This practice is currently utilized in our TBI population.
4. Undergoing therapeutic hypothermia with a target temperature under 35oC.
5. Known or prior history of severe TBI, intracranial hemorrhage or stroke that would interfere with cerebral oximetry (i.e. significant prior damage to the frontal lobes).
6. No current commitment to ongoing support by the medical team
7. Acute ST elevation myocardial infarction

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow | 6 hours
  mls/100g/min

IPD SHARING:
Plan to Share IPD: Undecided